CLINICAL TRIAL: NCT04105751
Title: Testing a Novel Manual Communication System for Mechanically Ventilated ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, J. Matthias Walz, Professor and Interim Chair, Dept of Anesthesiology and Perioperative Medicine, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H00010101
Record Dates: First submitted 2019-08-24; First posted 2019-09-26 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Communication; Ventilation Therapy; Complications
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Use of Device with post-use interview/questionnaire (Experimental): All patients will be asked to utilize device and will then be asked to provide feedback on their experiences. This may be done by interview or a questionnaire. There could be up to three sessions using the device. Each session is expected to last between 10 and 30 minutes. If the subject is interested in continuing, session could last up to one hour.
  Interventions: Device: Novel Communication System

INTERVENTIONS:
Device: Novel Communication System — Small hand held device that aids in answering questions. Used in conjunction with a tablet computer.

SUMMARY:
The objective of this study is to gather initial information about the testing of a novel manual communication system for mechanically ventilated Intensive Care Unit (ICU) subjects. This phase of the study is not hypotheses based; the goal is to gather data about which potential form factors and interaction modes of the proposed communication system are most intuitive for subjects and caregivers.

DETAILED DESCRIPTION:
Intensive Care Unit (ICU) admissions constitute a major part of hospital activity and resource allocation, and the number of patient days in ICUs and on mechanical ventilation is increasing. More than 5 million patients are admitted to an ICU annually in the United States, and approximately 55,000 critically ill patients are cared for each day. The most common cause for admission is respiratory insufficiency or failure; a study of data from 2005-2007 estimated that nearly 40 percent of ICU patients require mechanical ventilation.

Patients experience frequent emotional and psychiatric complications from ICU stays, including depression, anxiety, and post-traumatic stress disorder. One 2011 study found a prevalence of "clinically significant" depressive symptoms ranging from 17 percent to 43 percent among post-ICU patients. In 2013, it was reported that up to 50 percent of patients experience general anxiety symptoms one year after discharge, a rate much higher than in the broader US population.

Patients who temporarily lose the ability to speak report a high level of frustration. A study of 127 patients reported that, "two stressors, being intubated and not being able to talk, were significantly more stressful… than all the other stressors. The mean stressfulness score for [25] other stressors was between no distress and mild distress." Improving subject communication with ICU care team will likely require better technological interventions, and current best practice for assessing the optimal patient communication method is dependent on the evaluation of an experienced speech-language pathologist (SLP). Current approaches are insufficient for patient's needs, as one representative study described: "Patients rated 40% of the communication sessions with nurses as somewhat difficult to extremely difficult. Assistive communication strategies were uncommon, with little to no use of assistive communication materials (e.g., writing supplies, alphabet or word boards)." Designing an effective mode of communication for ICU patients unable to speak due to mechanical ventilation will likely improve patient's experiences and, potentially, long-term outcomes.

Some limited technologies exist to address these issues; however, they are not in widespread use due to a variety of reasons, including cost, lack of intuitiveness, and design that is not appropriate for the ICU setting. The investigators are designing a technological solution to assist ICU subjects in communicating with their caregivers, particularly nurses. The investigators are planning to do the initial testing of this device in the adult ICUs at the University of Massachusetts Memorial Medical Center at both the University Campus and Memorial Campus.

The purpose of this stage of the project is to test the current device and determine whether the physical factors and interaction modes that have been designed up to this point will be appropriate for the needs and desires of ICU subjects while communicating.

ELIGIBILITY:
Inclusion Criteria:

PHASE 1

1. Subjects who are awake, alert, and without clear evidence of delirium (GCS>13) adult subjects in the Memorial and University ICUs are eligible for this study.
2. Both subjects who are able to speak and subjects who are unable to speak (due to intubation or tracheostomy) will be sought to be included in the study.
3. Eligible subjects must have a history of being able to understand and communicate in written and spoken English or Spanish.
4. Any subject who is capable of consent but cannot speak will provide consent by signing the consent form if possible, with a witness, who is not a member of the research team, present who will sign the appropriate section of the consent form.

PHASE 2

1. Subjects who are awake with a GCS>10 (Motor 6, Verbal 1, Eye opening 3) adult subjects in the Memorial and University ICUs are eligible for this study.
2. Both subjects who are able to speak and subjects who are unable to speak (due to intubation or tracheostomy) will be sought to be included in the study.
3. Eligible subjects must have a history of being able to understand and communicate in written and spoken English or Spanish.
4. May enroll both adults capable of consent and cognitively impaired adults, who will provide assent, if possible, and will have consent given by their legally authorized representative.

Exclusion Criteria:

PHASE 1/PHASE 2

1. Spanish-speaking individuals may be included in the study under the following conditions:

   * Spanish interpreter is available in person or by phone for the consent process.
   * The consent process is followed as outlined in question 30-31, depending on whether subject is able to speak or not at this time.

   No other non-English-speaking subjects will be included in the study.
2. The following vulnerable populations will not be included in the study:

   * Pregnant women, non-adult individuals, prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Ability of user to make one or more selections in the software | 1 hour
  Whether the user is able to make one or more selections in the software will be evaluated.

SECONDARY OUTCOMES:
Duration of use | 1 hour
  The time spent using the system within a one-hour time frame will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: J. Matthias Walz, MD, Principal Investigator — UMass Medical School
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No